CLINICAL TRIAL: NCT00514163
Title: Randomized Phase II Study of Gemcitabine (GEM) Versus GEM+TS-1 for Advanced Pancreatic Cancer
Brief Title: GEM vs GEM+TS-1 for Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Clinical Cancer Research Organization (Other)
Responsible Party: Takaaki Ikari, Cancer Institute Ariake Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JACCRO PC-01
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic carcinoma; gemcitabine; S-1; phaseⅡstudy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): gemcitabine + S-1
  Interventions: Drug: gemcitabine + S-1
- 2 (Active Comparator): S-1
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: gemcitabine + S-1 — gemcitabine on day one and 8th S-1 po days 1 to14 every 3 weeks
  Other Names: gemzar; TS-1
  Arms: 1
Drug: gemcitabine — gemcitabine DIV on day one , 8th and 15th
  Other Names: gemzar
  Arms: 2

SUMMARY:
The primary objective of this study is to compare tumor response rate of the test arm(gemcitabine+S-1) with the control arm(gemcitabine alone) in patients with unresectable pancreatic cancer

DETAILED DESCRIPTION:
Pancreatic cancer is the fifth leading cause of cancer death in the United States. It is difficult to diagnose at its early stage and only 10-20% of patients are candidates for resection with 5-year survival rate of less than 10%. Patients with unresectable pancreatic cancer has a poor prognosis. Gemcitabine, a cytidine analogue, is the standard chemotherapeutic agent for the disease with median survival time(MST) ranging from 6 to 8 months. Phase Ⅲ study showed that combinations with other drugs, such as oxaliplatine or CDDP, did not contribute to survival time. TS-1, a new oral fluoropyrimidine which consists of the 5-FU prodrug tegafur (ftorafur, FT) and two enzyme inhibitors, CDHP (5-chloro-2,4-dihydroxypyridine) and OXO (potassium oxonate), in a molar ratio of 1(FT):0.4 (CDHP):1(OXO), is commercially available since late 90'in Japan. Phase II trials have demonstrated that S-1 was effective as a single agent for treatment of gastric (RR 44.6%), colorectal (RR 37.4%), head and neck, breast, non-small cell lung, and pancreatic cancers(20%). A combination of gemcitabine and TS-1 is found to be effective and promising in phase Ⅱ trial for metastatic pancreatic carcinoma in selected subjects, but the combination therapy has high rate of side effects. This phase Ⅱ randomized controlled study compares efficacy and feasibility of GEM+S-1 with GEM alone in patients with locally advanced and metastatic pancreatic cancer and performance status of 0-2, aiming at patients in rather ordinary clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven unresectable pancreatic carcinoma
2. There must be measurable lesions with multislice CT
3. ECOG Performance status 0-2
4. No other active cancer
5. No previous therapy such as radiotherapy, chemotherapy and immunotherapy
6. Adequate organ functions are preserved as WBC more than 4000/mm3,Hb more than 8.0g/dl,neutrophil more than 2000/mm3,platlet more than 100,000/mm3, AST less than 2.5 x normal or less than 5.0 x normal if the patient had known liver metastasis, bilirubin less than 2.0mg/dl, Ccr more than 60ml/min
7. No serious complications
8. Be able to eat food
9. Life expectancy of more than 8 weeks duration
10. Informed consent is obtained-

Exclusion Criteria:

1. Interstitial pneumonia
2. Uncontrollable diabetes, liver dysfunction, angina pectoris,or myocardial infarction with its onset within 3 months
3. Serious infection
4. Pregnant or lactating females
5. History of serious drug allergy
6. Serious other complications
7. Uncontrolled mental disorders -

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
response rate | during observation

SECONDARY OUTCOMES:
median survival time(MST) | during observation
time-to-progression(TTP) | from onset of regression to progression
toxicity | during observation
clinical benefit response | during observation

CONTACTS AND LOCATIONS:
Overall Officials: Takaaki Ikari, MD. PhD, Principal Investigator — Cancer Institute Ariake Hospital; Masafumi Suyama, M.D. PhD, Principal Investigator — Juntenndo University Hospital; Naoto Egawa, M.D. PhD, Principal Investigator — Komagome Hospital; Yasuji Omuro, M.D. PhD, Principal Investigator — Komagome Hospital; Takao Itoi, M.D. PhD, Principal Investigator — Tokyo Medical college; Atsushi Sofuni, M.D. PhD, Principal Investigator — Tokyo medical college
Locations (1):
- Cancer Institute Ariake Hospital, Tokyo, Japan